CLINICAL TRIAL: NCT01667341
Title: A Phase I/IIa, Randomized, Double-blind, Dose-ranging, Placebo-controlled Study of the Safety and Immunogenicity of a HSV-2 Vaccine Containing Matrix M-2 Adjuvant in Individuals With Documented Genital HSV-2 Genital Infection
Brief Title: Safety and Immunogenicity Study of Therapeutic HSV-2 Vaccine
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Genocea Biosciences, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: GEN-003-001
Record Dates: First submitted 2012-08-14; First posted 2012-08-17 (Estimated); Last update posted 2018-06-01 (Actual); Status verified 2018-05

CONDITIONS: Genital Herpes Simplex Type 2
Keywords: HSV; Herpes; genital infection; vaccine
MeSH Terms: conditions — Herpes Simplex

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (7):
- Low Dose GEN-003 with Matrix M-2 (Experimental): 10µg GEN-003, 50µg Matrix M-2 Adjuvant
  Interventions: Biological: GEN-003 with Matrix M-2
- Mid Dose GEN-003 with Matrix M-2 (Experimental): 30µg GEN-003, 50µg Matrix M-2 Adjuvant
  Interventions: Biological: GEN-003 with Matrix M-2
- High Dose GEN-003 with Matrix M-2 (Experimental): 100µg GEN-003, 50µg Matrix M-2 Adjuvant
  Interventions: Biological: GEN-003 with Matrix M-2
- Low Dose GEN-003 Only (Experimental): 10µg GEN-003
  Interventions: Biological: GEN-003
- Mid Dose GEN-003 Only (Experimental): 30µg GEN-003
  Interventions: Biological: GEN-003
- High Dose GEN-003 Only (Experimental): 100µg GEN-003
  Interventions: Biological: GEN-003
- Placebo (Placebo Comparator): 0.5 mL phosphate buffered saline
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: GEN-003 with Matrix M-2 — IM administration of GEN-003 Vaccine with 50ug Matrix M-2 Adjuvant.
  Arms: High Dose GEN-003 with Matrix M-2; Low Dose GEN-003 with Matrix M-2; Mid Dose GEN-003 with Matrix M-2
Biological: GEN-003 — IM administration of GEN-003 Vaccine, antigens alone (without adjuvant).
  Arms: High Dose GEN-003 Only; Low Dose GEN-003 Only; Mid Dose GEN-003 Only
Biological: Placebo — IM administration of 0.5 mL dose of Dulbecco's phosphate buffered saline.
  Other Names: PBS; DPBS
  Arms: Placebo

SUMMARY:
Randomized, double-blind, placebo-controlled, dose escalation study. There will be 3 cohorts of patients defined by the antigen dose (10, 30 or 100 µg of each antigen), and within each cohort, patients will be randomized at a ratio of 3:1:1 to one of the following:

1. GEN-003/M2: GEN-003 plus Matrix M-2 adjuvant (50 µg per dose)
2. GEN-003: Antigens alone
3. Placebo (DPBS diluent)

Each Cohort is divided into 2 Groups. For each dose cohort, immunizations begin with a Pilot Group. Immunization of the remainder of the Group "Continuation Group") is contingent upon successful review of data from the Pilot Group through Day 7 after immunization. Dose escalation to the next dose level Cohort proceeds after evaluation of safety data from all patients in the prior Cohort and only after all specified safety criteria are met. The total numbers of patients in each Group and Cohort are as follows:

* 10 µg Cohort: 10 Pilot Group, 40 Continuation Group (50 Total)
* 30 µg Cohort: 10 Pilot Group, 40 Continuation Group (50 Total)
* 100 µg Cohort: 10 Pilot Group, 40 Continuation Group (50 Total)
* Totals per group: 30 Pilot Group, 120 Continuation Group (150 Total Patients)

Subjects will receive 3 doses of the assigned treatment (GEN-003/M-2, GEN-003, or placebo) at 3 week intervals. Sampling from mucocutaneous genital sites for viral shedding will be done twice daily for 28 days prior to the first immunization (baseline shedding), and again following the last immunization. Follow-up for safety monitoring will be conducted for 12 months after the last immunization.

ELIGIBILITY:
Inclusion Criteria:

* Men and women ages 18 to 50 years, inclusive.
* Willing to practice a highly effective method of contraception that includes the use of a barrier method such as a condom.
* Diagnosis of genital HSV-2 infection for > 1 year supported by ONE of the following documented in the medical history or performed at screening:

  * Western blot for HSV-2
  * Type-specific polymerase chain reaction (PCR) or viral culture
  * Compatible clinical history AND HSV-2 ELISA (HerpSelect) index value >3.5
* A history of at least 3 and no more than 9 reported clinical occurrences in the prior 12 months, or, if currently on suppressive therapy, history of at least 3 and no more than 9 reported clinical occurrences in the 12 months prior to initiation suppressive therapy.
* Good general health status as determined by screening evaluation completed within 90 days prior to immunization. Any out of range screening clinical laboratory values should be considered not clinically significant by the Investigator.
* Patient has provided written informed consent.
* Ability and willingness to perform and comply with all study procedures including attending clinic visits as scheduled. Note: patients must provide, by the day of randomization, a minimum of 28 (equivalent of 14 days) baseline viral swab samples to continue to be eligible and be randomized).

Exclusion Criteria:

* On suppressive antiviral medication within 7 days of baseline viral shedding evaluation.
* Immunocompromised individuals, including those receiving systemic corticosteroids or other immunosuppressive agents.
* Positive serologic test for HIV-1 infection; positive hepatitis B surface antigen (HBsAg) or antibody for hepatitis C (anti-HCV).
* Active lesions consistent with herpetic disease at the time of scheduled immunization.
* Pregnant or nursing women.
* Receipt of any investigational drug within 30 days of the first scheduled day of immunization.
* History of hypersensitivity to any component of the vaccine.
* History of genital HSV-1 infection.
* History of: (1) any form of ocular HSV infection, (2) HSV-related erythema multiforme, or (3) herpes meningitis or encephalitis.
* Any other condition which in the opinion of the Investigator would interfere with the successful completion of the study protocol.
* History of drug or alcohol abuse that, in the opinion of the Investigator, would interfere with the patient's ability to comply with the requirements of the study.
* Prior immunization with a vaccine containing HSV-2 antigens.
* Receipt of blood products within 90 days of the first immunization.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 143 (Actual)
Dates: Start 2012-07 (Actual); Primary Completion 2014-05-09 (Actual); Study Completion 2014-05-09 (Actual)

PRIMARY OUTCOMES:
Number of patients with adverse events as a measure of safety and tolerability | 57 Weeks

SECONDARY OUTCOMES:
Immunogenicity measured by humoral (antibody) and T-cell responses to vaccine antigens | 33 weeks
Change in proportion of days with detectable viral shedding | 6 weeks

CONTACTS AND LOCATIONS:
Locations (7):
- United States (7):
  - University of Alabama Vaccine Research Unit, Birmingham, Alabama
  - Indiana University Infectious Disease Research, Indianapolis, Indiana
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Westover Heights Clinic, Portland, Oregon
  - Center for Clinical Studies - Houston, Houston, Texas
  - Center for Clinical Studies - Clear Lake/Webster, Webster, Texas
  - UW Virology Research Clinic, Seattle, Washington

REFERENCES:
- [Derived] Bernstein DI, Wald A, Warren T, Fife K, Tyring S, Lee P, Van Wagoner N, Magaret A, Flechtner JB, Tasker S, Chan J, Morris A, Hetherington S. Therapeutic Vaccine for Genital Herpes Simplex Virus-2 Infection: Findings From a Randomized Trial. J Infect Dis. 2017 Mar 15;215(6):856-864. doi: 10.1093/infdis/jix004. PMID 28329211